CLINICAL TRIAL: NCT02033070
Title: Single Center Patient Registry Using Radio Frequency Ablation of Barrett's Esophagus Using HALO System
Brief Title: Patient Registry: Radio Frequency Ablation of Barrett's Esophagus Using HALO System
Acronym: HALO
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Ochsner Health System (Other)
Responsible Party: Principal Investigator, Virendra Joshi, Virendra Joshi, MD, Ochsner Health System
Other Study IDs: Barrett's RFA
Record Dates: First submitted 2014-01-08; First posted 2014-01-10 (Estimated); Last update posted 2014-01-10 (Estimated); Status verified 2014-01

CONDITIONS: Barrett's Esophagus
Keywords: RFA
MeSH Terms: conditions — Barrett Esophagus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples Without DNA — Serum from Biopsy
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Non-Dysplastic IM, LGD, HGD

SUMMARY:
The purpose of this study is to provide a tool for physicians to compare outcome data related to the use of the HALO Ablation Systems. This study is a single-center patient registry which will contribute to a framework for treatment and follow-up of patients with Barrett's Esophagus.

ELIGIBILITY:
Inclusion Criteria:

* candidate for ablation of Barrett's Esophagus with the HALO Ablation System (Prospective)
* received an ablation with the HALO Ablation System to treat Barrett's Esophagus (Retrospective)
* candidate agrees to proposed follow-up schedule of yearly surveillance following treatment
* signs consent

Exclusion Criteria:

* has not been diagnosed with Barrett's Esophagus

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Adult patients presenting with esophageal intestinal metaplasia (IM), including the pathological subclasses of non-dysplastic IM, low-grade dysplasia (LGD) and high-grade dysplasia (HGD)
Sampling Method: Non-Probability Sample
Dates: Start 2013-11; Primary Completion 2015-11 (Estimated)

PRIMARY OUTCOMES:
Endoscopic clearance rate for Barrett's Esophagus | Outcome measure is assessed at Month 12

SECONDARY OUTCOMES:
Histological clearance rate for intestinal metaplasia | Biopsy taken at 12 months

OTHER OUTCOMES:
Histological clearance rate for dysplasia | Biopsy taken at 12 months to determine effectiveness

CONTACTS AND LOCATIONS:
Overall Officials: Virendra Joshi, MD, Principal Investigator — Oshsner Clinic Foundation and Medical Center-Kenner
Locations (1):
- Ochsner Medical Center, Kenner, Louisiana, United States